CLINICAL TRIAL: NCT03564821
Title: A Phase 1 Study of IDH1 Inhibition Using Ivosidenib as Maintenance Therapy for IDH1-mutant Myeloid Neoplasms Following Allogeneic Stem Cell Transplantation
Brief Title: IDH1 Inhibition Using Ivosidenib as Maintenance Therapy for IDH1-mutant Myeloid Neoplasms Following Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Amir Fathi, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-123
Record Dates: First submitted 2018-06-07; First posted 2018-06-21 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: IDH1 Mutation Myeloid Neoplasms
Keywords: myeloid neoplasms
MeSH Terms: interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ivosidenib (500mg/day) (Experimental): -Ivosidenib will be administered orally every day
  Interventions: Drug: Ivosidenib
- Ivosidenib (250mg/day) (Experimental): -Ivosidenib will be administered orally every day
  Interventions: Drug: Ivosidenib

INTERVENTIONS:
Drug: Ivosidenib — Ivosidenib is an inhibitor of the protein IDH1

SUMMARY:
This research study is studying a drug as a possible treatment for IDH1-mutant myeloid neoplasms.

-The drug involved in this study is ivosidenib (AG-120)

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved ivosidenib as a treatment for any disease.

Ivosidenib is an inhibitor of the protein IDH1. Ivosidenib is currently being studied as a treatment for myeloid cancers like acute myeloid leukemia or myelodysplastic syndromes with an IDH1 mutation. This study is examining whether or not ivosidenib is beneficial and well-tolerated as an agent to prevent the relapse of IDH1-mutated acute myeloid leukemia or other myeloid neoplasms after hematopoietic stem cell transplantation. IDH1 is an enzyme that, when mutated, can overproduce metabolites (substances that help with metabolism) and compounds that contribute to the growth of tumors and cancerous cells. Ivosidenib may help block the over production of these substances and possibly reduce the chances of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of IDH1(R132)-mutant acute myeloid leukemia (AML), myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML). IDH1 mutations could have been detected by any mutational technique at any prior point including at diagnosis or remission.
* Between the ages of 18 and 75 years
* Will undergo allogeneic hematopoietic stem cell transplantation (HSCT) for their malignancy. Conditioning may be either conventional myeloablative (MAC) or reduced intensity conditioning (RIC).
* HSCT Donor will be one of the following:

  * 5/6 or 6/6 (HLA-A, B, DR) matched related donor
  * 7/8 or 8/8 (HLA-A, B, DR, C) matched unrelated donor. Matching in the unrelated setting must be at the allele level.
  * Haploidentical related donor, defined as ≥ 3/6 (HLA-A, B, DR) matched --≥ 4/6 (HLA-A, B, DR) umbilical cord blood (UCB). Matching in the UCB setting is at the antigen level. Recipients may receive either one or two UCB units. In the case of 2 UCB units, both units must have been at least 4/6 matched with the recipient.
* ECOG performance status ≤ 2
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1000/µL without growth factor support (e.g. GCSF) in the previous 7 days
  * Platelet count ≥ 50,000/µL without transfusional support in the previous 7 days
  * AST (SGOT), ALT (SGPT) and Alkaline phosphatase < 3x institutional upper limit of normal (ULN)
  * Direct bilirubin < 2.0 mg/dL
  * Calculated creatinine clearance ≥ 40 mL/min (Cockcroft-Gault formula)
  * LVEF must be equal to or greater than 40%, as measured by MUGA scan or echocardiogram
* Female patients of childbearing potential must have a negative pregnancy test
* The effects of ivosidenib on the developing human fetus are unknown. For this reason female participants of child-bearing potential and male participants must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) during the entire study treatment period and through 90 days after the last dose of treatment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplants.
* Evidence of relapsed/recurrent/residual disease as assessed by bone marrow aspirate and biopsy performed within 42 days prior to study entry.
* History of other malignancy(ies) unless

  * the participant has been disease-free for at least 5 years and is deemed by the investigator to be at low risk of recurrence of that malignancy, or
  * the only prior malignancy was cervical cancer in situ and/or basal cell or squamous cell carcinoma of the skin
* Known diagnosis of active hepatitis B or hepatitis C
* Current or history of congestive heart failure New York Heart Association (NHYA) class 3 or 4, or any history of documented diastolic or systolic dysfunction (LVEF < 40%, as measured by MUGA scan or echocardiogram)
* Current or history of ventricular or life-threatening arrhythmias or diagnosis of long-QT syndrome
* QTc interval (i.e., Friderica's correction [QTcF]) ≥ 450 ms or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) at screening
* Systemic infection requiring IV antibiotic therapy within 7 days preceding the first dose of study drug, or other severe infection
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with study drug. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28 Days
  Participants will be enrolled in standard 3 + 3 dose escalation cohorts in order to determine the maximum tolerated dose (MTD). The first 3 participants will be started on 500mg of Ivosidenib, administered daily for 28 consecutive days (1 cycle). If the 500mg/day dose level is tolerated, an additional 10 participants will be treated at this dose level. If the 500mg/day dose is not tolerated, the dose will be decreased to 250mg/day. If 250mg daily is tolerated, then an additional 10 participants will be treated at 250mg daily. The only doses studied will be 500mg daily and 250mg daily (the latter, if necessary). If 250mg daily dosing is not tolerated, then the study will end without expansion. Dose limiting toxicities are assessed and graded using Common Terminology Criteria for Adverse Events (CTCAE 4).

SECONDARY OUTCOMES:
Ivosidenib-related Adverse Events, categorized by grade | From the start of treatment until 30 days after the end of treatment, up to 13 months total
  Adverse events will be assessed and graded using Common Terminology Criteria for Adverse Events (CTCAE 4).
Cumulative incidence of acute GVHD | From the start of treatment with Ivosidenib until the onset of Acute GVHD, up to 100 days
  Cumulative incidence of acute graft versus host disease (GVHD), measured from start of treatment with Ivosidenib.
Cumulative incidence of chronic GVHD | From the start of treatment with Ivosidenib until the onset of chronic GVHD, up to 24 months
  The cumulative incidence of chronic GVHD, measured from start of treatment with Ivosidenib. Chronic GVHD will be assessed using the National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease.
Plasma and marrow 2-hydroxyglutarate levels | Screening, cycle 1 days 8 and 15 (cycles are 28 days), before the start of cycles 2 and 3, and at the time of relapse; up 24 months total time
IDH clonal evolution and mutational burden | Screening, cycle 1 days 8 and 15 (cycles are 28 days), before the start of cycles 2 and 3, and at the time of relapse; up 24 months total time
  Isocitrate dehydrogenase (IDH) clonal evolution and mutational burden in patients with IDH1-mutant myeloid neoplasms who receive Ivosidenib after hematopoietic stem cell transplantation. Next-generation sequencing will be used to assess mutational burden (i.e. the fraction of AML cells harboring IDH mutations, corrected for copy number) at various time points. SNaPshot genotyping analysis platform will be used to perform these analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Amir T Fathi, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Johns Hopkins Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shallis RM, Podoltsev NA. Maintenance therapy for acute myeloid leukemia: sustaining the pursuit for sustained remission. Curr Opin Hematol. 2021 Mar 1;28(2):110-121. doi: 10.1097/MOH.0000000000000637. PMID 33394722

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT03564821/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT03564821/ICF_001.pdf